CLINICAL TRIAL: NCT01700530
Title: Exercise, Statins, and the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: University of Missouri-Columbia (Other); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09CRP2260136
Record Dates: First submitted 2012-09-26; First posted 2012-10-04 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Metabolic Syndrome; Obese; Sedentary
Keywords: mitochondria; fitness; statins; cholesterol; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Sedentary Behavior | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Simvastatin; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Statin (Experimental): Statins (40mg/day)for an average of 12 weeks
  Interventions: Drug: Statin
- Exercise only (Experimental): 12 weeks of exercise training (5 days a week for 45-50 min a session)
  Interventions: Other: Exercise only
- Statins + Exercise (Active Comparator): Statins (40mg/day of simvastatin) plus exercise training (5 days/wk) for 12 weeks
  Interventions: Other: Statins + Exercise

INTERVENTIONS:
Drug: Statin — Statins (40mg/day)for 12 weeks
  Other Names: simvastatin
  Arms: Statin
Other: Exercise only — 12 weeks of exercise training (5 days a week for 45-50 min a session)
  Other Names: Physical activity
  Arms: Exercise only
Other: Statins + Exercise — Statins (40mg/day of simvastatin) plus exercise training (5 days/wk for 45-50 min a session) for 12 weeks
  Other Names: Statins + Physical Activity
  Arms: Statins + Exercise

SUMMARY:
Here we tested if statins or exercise plus statins had a greater capacity to lower metabolic syndrome risk factors in sedentary individuals with at least 2 metabolic syndrome risk factors. We also examined if statins impacted exercise response for mitochondrial content in muscle or aerobic fitness.

DETAILED DESCRIPTION:
OBJECTIVES: Determine if simvastatin impairs exercise training adaptations.

BACKGROUND: Statins are commonly prescribed in combination with therapeutic lifestyle changes, including exercise, to reduce cardiovascular disease risk in patients with the metabolic syndrome. Statin use has been linked to skeletal muscle myopathy and impaired mitochondrial function, but it is unclear whether statin use alters adaptations to exercise training.

METHODS: We examined the effects of simvastatin on changes in cardiorespiratory fitness and skeletal muscle mitochondrial content in response to aerobic exercise training. Sedentary overweight or obese adults with at least 2 metabolic syndrome risk factors (defined according to National Cholesterol Education Panel Adult Treatment Panel III criteria) were randomized to 12 weeks of aerobic exercise training or to exercise in combination with simvastatin (40 mg per day). The primary outcomes were cardiorespiratory fitness and skeletal muscle (vastus lateralis) mitochondrial content (citrate synthase enzyme activity).

ELIGIBILITY:
Inclusion Criteria:

* Sedentary metabolic syndrome subjects will be 25-59 y of age
* overweight to Class I or II obese (BMI 25-39 kg/m2) men and women
* 2 of 4 other characteristics of the metabolic syndrome including fasting glucose of 100 to 125 mg/dl; waist circumference greater than 102 cm in men and 88 cm in women, serum triglyceride concentration greater than 150 mg/dl, HDL-C concentrations less than 40 mg/dl in men and 50 mg/dl in women, and blood pressure greater than 130/85 mmHG
* Women must be taking birth control or be postmenopausal.

Exclusion Criteria:

* Diagnosed cardiovascular disease or diabetes or disease
* Symptoms that could alter their ability to perform exercise
* Fasting blood glucose of greater than 126 mg/dl
* Smoking
* Taking any medications or supplements (e.g., statins, fibrates, metformin, thiazolidenediones, anti-hypertensives (ACE-inhibitors and angiotensin blockers) which could affect blood lipids or insulin sensitivity.
* Women who are pregnant or plan to become pregnant during the duration of the study
* Individuals exercising regularly (more than one 30 min session per week)
* Individuals with an orthopedic limitations for walking.
* Report any allergies to the medications (statins, lidocaine)

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2007-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Thyfault, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

REFERENCES:
- [Derived] Mikus CR, Boyle LJ, Borengasser SJ, Oberlin DJ, Naples SP, Fletcher J, Meers GM, Ruebel M, Laughlin MH, Dellsperger KC, Fadel PJ, Thyfault JP. Simvastatin impairs exercise training adaptations. J Am Coll Cardiol. 2013 Aug 20;62(8):709-14. doi: 10.1016/j.jacc.2013.02.074. Epub 2013 Apr 10. PMID 23583255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: If meeting qualifications after initial phone screening, subject consented followed by another round of screening to determine if they had 2/5 risk factors or not which eliminated many subjects. Thus the difference between the 121 subjects reported for who signed consents and the 50 who entered the participant flow module.
Period: Overall Study
Arm/Group | Statin | Exercise Only | Statins + Exercise
Started | 9 | 21 | 20
Completed | 9 | 18 | 19
Not Completed | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Sedentary, obese, 2/5 metabolic syndrome risk factors, males and females
Groups:
- Total: Total of all reporting groups
Arm/Group | Statin | Exercise Only | Statins + Exercise | Total
Number analyzed (Participants) | 9 | 21 | 20 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (10) | 44 (12) | 43 (9) | 44 (10)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 21 | 20 | 50
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 13 | 11 | 28
  Male | 5 | 8 | 9 | 22
Region of Enrollment [Number; unit: participants]
  United States | 9 | 21 | 20 | 50

OUTCOME MEASURES:

1. Primary Outcome: % Change in VO2max (Fitness)
Description: % change in fitness between baseline and after 12 weeks of treatment will be assessed by VO2max
Time Frame: Change from Baseline to 12 weeks
Population: Statins blocked exercise induced change in fitness
Measure: Mean (Standard Deviation); unit: percentage change of VO2max
Arm/Group | Statin | Exercise Only | Statins + Exercise
Number analyzed (Participants) | 9 | 18 | 19
percentage change of VO2max | 0 (6) | 10 (5) | 1.5 (6)
Statistical Analysis 1: Comparison: Statin vs Exercise Only vs Statins + Exercise; Test type: Superiority or Other; p < 0.05, ANOVA

2. Secondary Outcome: Skeletal Muscle Mitochondrial Content (Citrate Synthase Enzyme Activity)
Description: % change in skeletal muscle mitochondrial content (measured by citrate synthase enzyme activity) from pre to post intervention
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Statin | Exercise Only | Statins + Exercise
Number analyzed (Participants) | 9 | 19 | 18
percent change | 0 (10) | 13 (7) | -4.5 (8)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Statin | Exercise Only | Statins + Exercise
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/9 | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No